CLINICAL TRIAL: NCT03295409
Title: Testing Familial Self-affirmation for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Christopher Armitage, Professor of Health Psychology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Chun_1
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Standard self-affirmation (Experimental): Participants are asked to form a self-affirming implementation intention at the end of a questionnaire:
  The beginning to a sentence appears below. Below it are 4 different ways of completing the sentence. On the lines below, please write out the beginning of the sentence and then complete it with 1 of the 4 options we have given you.
  If I feel threatened or anxious, then I will…
  * think about the things I value about myself
  * remember things that I have succeeded in
  * think about what I stand for
  * think about things that are important to me
  If…___________________________________________________________________
  Interventions: Behavioral: Self-affirmation
- Experimental: Familial self-affirmation (Experimental): Participants are asked to form a self-affirming implementation intention at the end of a questionnaire:
  The beginning to a sentence appears below. Below it are 4 different ways of completing the sentence. On the lines below, please write out the beginning of the sentence and then complete it with 1 of the 4 options we have given you.
  If I feel threatened or anxious, then I will…
  * think about the things my family and I value about ourselves
  * remember things that my family and I have succeeded in
  * think about what my family and I stand for
  * think about things that are important to my family and me
  If…__________________________________________________________________
  Interventions: Behavioral: Self-affirmation
- Control (No Intervention): Participants are asked to complete a questionnaire.

INTERVENTIONS:
Behavioral: Self-affirmation — Participants are asked to complete a standard questionnaire and on the last page they are asked to form a self-affirming implementation intention by copying out a sentence.
  Arms: Experimental: Familial self-affirmation; Experimental: Standard self-affirmation

SUMMARY:
Evidence suggests that affirming the self can help people to make changes in their health behavior. Typically, people affirm a personally-important value, but evidence suggests that affirming the values of family ("familial self-affirmation") might exert stronger effects. The aim of the present study is to examine the effects of familial self-affirmation versus standard self-affirmation versus a control group on smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Smoker

Exclusion Criteria:

* Non-smoker
* Unable or unwilling to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 1 month
  Self-reported quitting
Quit attempts | 1 month
  Self-reported quit attempts
Nicotine dependence | 1 month
  Self-reported nicotine dependence
Craving | 1 month
  Self-reported cravings

SECONDARY OUTCOMES:
Habit | 1 month
  Self-reported habit
Self-regulation | 1 month
  Self-reported self-regulation
Subjective well-being | 1 month
  Self-reported subjective well-being

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - HC Engineering Company, Hong Kong
  - Perfect Match Wedding Service, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised SPSS file